CLINICAL TRIAL: NCT05252182
Title: Comprehensive Geriatric Assessment in the Emergency Department: a Prospective Cohort Study of Clinical and Process Outcomes
Brief Title: Comprehensive Geriatric Assessment in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Limerick (Other)
Collaborators: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, IDE O SHAUGHNESSY, Principal Investigator, University of Limerick
Other Study IDs: ED-CGA
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Frailty
Keywords: older adults; frailty; emergency department; comprehensive geriatric assessment
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comprehensive geriatric assessment (CGA) has been shown to improve outcomes in an inpatient setting; however, there is currently no compelling evidence of benefit for CGA interventions within the Emergency Department (ED). This study aims to explore the clinical and process outcomes of older adults who receive interdisciplinary ED-CGA over a period of six months after their initial ED attendance.

DETAILED DESCRIPTION:
The significant growth in ED attendances is a growing public health issue, with attendances by older adults accelerating over the past decade, beyond that due to population ageing alone. The reasons underlying older adults higher rate of healthcare utilisation, specifically ED usage, are multifaceted. However, the most potent intrinsic factor is the clinical condition of frailty. The presence of diminished homeostatic reserves leaves older adults more susceptible to acute exacerbations of comorbid and long-term conditions, which result in a concomitant increased demand for emergency care.

A presentation to an ED can be viewed as a sentinel event for an older adult. Conversely, it affords clinicians an opportunity to identify a high risk cohort followed by delivery of a holistic and bio-psychosocial intervention to mitigate against suboptimal outcomes. CGA is considered the gold standard approach to improving a range of outcomes for frail older adults in acute hospitals. Research has demonstrated that it is feasible to embed CGA within the ED and a model of care delivered by interdisciplinary teams incorporating geriatric competencies into their service has been recommended to meet the emergency and urgent care needs of this patient population within the ED. Despite this recommendation, there is no compelling evidence that ED-CGAs are clinically effective at improving clinical and process outcomes.

An ED based interdisciplinary team aim to improve the quality of care and outcomes of older adults through delivery of a CGA. CGA is an intensive interdisciplinary intervention, which assesses an older adult in a holistic fashion incorporating medical, functional, physical and psychological process of care. The team compromises a senior registrar in Geriatric Medicine, specialist geriatric nurse, senior occupational therapist, senior physiotherapist, and senior medical social worker. The investigators propose to explore the clinical and process outcomes of older adults who receive an interdisciplinary ED-CGA over a period of six months after their initial ED attendance through the conduct of a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years;
* Identification of Seniors at Risk score of ≥ 2;
* Manchester Triage System category of 2 to 5;
* Presenting with a medical complaint.

Exclusion Criteria:

* Older adults who are deemed not to have capacity to provide informed consent;
* Older adults who present to the ED outside of the operational working hours (Monday-Friday, 08:00-16:00) of the interdisciplinary ED-CGA team;
* Older adults presenting with acute cardiac and/or neurological pathology;
* Older adults presenting with injuries that require surgical intervention;
* Older adults presenting with high illness acuity, which necessitates treatment in the resuscitation room for the duration of their ED stay.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Older adults aged ≥ 65 years who screen positive for risk of adverse outcomes following ED attendance.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of hospital admission from the ED index attendance. | 6 months
  Number of participants who are admitted to hospital following their index ED attendance

SECONDARY OUTCOMES:
Incidence of functional decline (including functional decline at discharge from hospital among the cohort admitted from the ED). | 30 days and 6 months
  Functional decline is defined as a net decrease in the number of activities of daily living performed independently as measured by the self-reported Barthel Index. The sum score of all subscales may range from 0-20 points, where 0 indicates the maximum level of dependency and 20 indicates maximum independence.
Patient satisfaction with the ED index attendance | 30-day follow-up
  Participants will rate their satisfaction across a number of domains using the 18-item Patient Satisfaction Questionnaire. The sum score of all subscales may range from 18 to 90 points, where 18 points is the poorest possible evaluation and 90 points the best.
Number of unscheduled ED re-attendances | 30 days and 6 months
  Number of participants who experienced an unscheduled ED re-attendance following their index attendance
Number of unscheduled hospital admissions | 30 days and 6 months
  Number of participants who experienced an unscheduled hospital (re)admission following their ED index attendance
Nursing home admission | 30 days and 6 months
  Number of participants who were admitted to a nursing home or residential care facility following their ED index attendance
Mortality | 30 days and 6 months
  Number of participants who died following their ED index attendance
Healthcare utilisation | 30 days and 6 months
  Number and duration of services that participants were in receipt of following ED index attendance e.g. specialist geriatric ambulatory care hub attendances, GP visits, public health nurse visits, home care support, outpatient clinic attendance, health and social care professionals input etc.

CONTACTS AND LOCATIONS:
Overall Officials: Íde O'Shaughnessy, MSc, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] McCusker J, Bellavance F, Cardin S, Trepanier S, Verdon J, Ardman O. Detection of older people at increased risk of adverse health outcomes after an emergency visit: the ISAR screening tool. J Am Geriatr Soc. 1999 Oct;47(10):1229-37. doi: 10.1111/j.1532-5415.1999.tb05204.x. PMID 10522957
- [Background] Mackway-Jones K ed: Emergency triage. London: BMJ Publishing Group. 1997.
- [Background] Marshall GN, Hays RD: The Patient Satisfaction Questionnaire Short Form (PSQ-18). Santa Monica, CA: Rand; 1994.
- [Background] Conroy SP, Turpin S. New horizons: urgent care for older people with frailty. Age Ageing. 2016 Sep;45(5):577-84. doi: 10.1093/ageing/afw135. Epub 2016 Aug 1. PMID 27496917
- [Background] Morley C, Unwin M, Peterson GM, Stankovich J, Kinsman L. Emergency department crowding: A systematic review of causes, consequences and solutions. PLoS One. 2018 Aug 30;13(8):e0203316. doi: 10.1371/journal.pone.0203316. eCollection 2018. PMID 30161242
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Lowthian JA, McGinnes RA, Brand CA, Barker AL, Cameron PA. Discharging older patients from the emergency department effectively: a systematic review and meta-analysis. Age Ageing. 2015 Sep;44(5):761-70. doi: 10.1093/ageing/afv102. Epub 2015 Aug 10. PMID 26265674
- [Background] Sanders AB, Witzke D, Jones JS, et al.: Principles of care and application of the geriatric emergency care model. In: Sanders AB, ed. Emergency Care of the Elder Person. St Louis: Beverly Cracom Publications, 1996; 59-93.
- [Background] Vermeiren S, Vella-Azzopardi R, Beckwee D, Habbig AK, Scafoglieri A, Jansen B, Bautmans I; Gerontopole Brussels Study group. Frailty and the Prediction of Negative Health Outcomes: A Meta-Analysis. J Am Med Dir Assoc. 2016 Dec 1;17(12):1163.e1-1163.e17. doi: 10.1016/j.jamda.2016.09.010. PMID 27886869
- [Background] Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, Conroy SP, Kircher T, Somme D, Saltvedt I, Wald H, O'Neill D, Robinson D, Shepperd S. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD006211. doi: 10.1002/14651858.CD006211.pub3. PMID 28898390
- [Background] Conroy SP, Stevens T, Parker SG, Gladman JR. A systematic review of comprehensive geriatric assessment to improve outcomes for frail older people being rapidly discharged from acute hospital: 'interface geriatrics'. Age Ageing. 2011 Jul;40(4):436-43. doi: 10.1093/ageing/afr060. Epub 2011 May 26. PMID 21616954
- [Background] Conroy SP, Ansari K, Williams M, Laithwaite E, Teasdale B, Dawson J, Mason S, Banerjee J. A controlled evaluation of comprehensive geriatric assessment in the emergency department: the 'Emergency Frailty Unit'. Age Ageing. 2014 Jan;43(1):109-14. doi: 10.1093/ageing/aft087. Epub 2013 Jul 23. PMID 23880143
- [Background] Harding S. Comprehensive geriatric assessment in the emergency department. Age Ageing. 2020 Oct 23;49(6):936-938. doi: 10.1093/ageing/afaa059. PMID 32315396
- [Derived] O'Shaughnessy I, Robinson K, O'Connor M, Conneely M, Steed F, Ryan D, Carey L, Shchetkovsky D, Shanahan E, Leahy A, Quinn C, Sheikhi A, Galvin R. Comprehensive geriatric assessment in the emergency department: A protocol for a prospective cohort study. HRB Open Res. 2022 Sep 14;5:26. doi: 10.12688/hrbopenres.13504.2. eCollection 2022. PMID 36313054